CLINICAL TRIAL: NCT04816240
Title: Evaluation of Albumin and Midodrine Versus Albumin Alone in Outcome of Refractory Ascites in Patients With Decompensated Cirrhosis - A Double Blind Randomized Controlled Trial."
Brief Title: Evaluation of Albumin and Midodrine Versus Albumin Alone in Outcome of Refractory Ascites in Patients With Decompensated Cirrhosis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-40
Record Dates: First submitted 2021-03-15; First posted 2021-03-25 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-03

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Midodrine; Albumins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midodrine + Albumin +Standard Medical Treatment (Experimental): SMT + Albumin + Midodrine (5mg thrice daily and will be increased every 3 days upto 15 mg thrice daily with target MAP (>75 mm and <90).
  Interventions: Drug: Midodrine; Biological: Albumin; Other: Standard Medical Treatment
- Albumin + Standard Medical Treatment+ Placebo (Active Comparator): 80grams/week for 2 weeks followed by 40gram/week + Placebo
  Interventions: Biological: Albumin; Other: Standard Medical Treatment; Other: Placebo

INTERVENTIONS:
Drug: Midodrine — 5mg thrice daily and will be increased every 3 days upto 15 mg thrice daily with target MAP (>75 mm and <90)
  Arms: Midodrine + Albumin +Standard Medical Treatment
Biological: Albumin — 80grams/week for 2 weeks followed by 40gram/week
Other: Standard Medical Treatment — Standard Medical Treatment
Other: Placebo — Placebo
  Arms: Albumin + Standard Medical Treatment+ Placebo

SUMMARY:
The project is about evaluation of albumin and midodrine versus albumin alone in outcome of refractory ascites in patients with decompensated cirrhosis.

Cirrhosis is a leading cause of disability and mortality worldwide. Cirrhosis occurs in 50% of patients over 10 years. Decompensated cirrhosis carries a poor prognosis because the median survival time is about 2 years and it imposes a heavy burden on health care costs mainly due to the need for repeated hospital admission. The mortality is approximately 40% at 1 year and 50% at 2 years (12.7 per 100,000 population). A lot of times the prognosis is poor and the main factors leading to it are - AKI/HRS-NAKI, Hyponatremia, Grade of ascites-Refractory ascites, Sarcopenia, low Mean arterial pressure.

Post review of the literature, it is realized that there are some gap areas -

* It is unknown whether combination of vasoconstrictor with albumin further decreases the need for paracentesis in patients of refractory ascites.
* There are no studies till date on using combination of vasoconstrictor with albumin for refractory ascites.
* There are no studies evaluating the prevalence and incidence of HRS-NAKI using the new definitions in patients with refractory ascites and impact of combining vasoconstrictor and albumin in improving renal outcomes in these patients.

DETAILED DESCRIPTION:
Study population All patients with decompensated cirrhosis with refractory ascites who get admitted under the Department of Hepatology at Institute of Liver and Biliary Sciences, who fulfilthe inclusion criteria, exclusion criteria and provide informed consent

* Study design Single Centre Placebo Controlled an open level Randomised Controlled Trial
* Study period 1 year from ethics approval.
* Sample size Assuming that survival rate with albumin and midodrine is 80%, whereas with albumin alone is 60% ( ie. 20% absolute difference is observed with alpha of 5% power so we need to enroll 170 cases allotted in 2 groups further taking 10% as dropout rate. It was decided to enroll 200 cases allotted in 2 groups randomly by block randomization method taking block size as 10
* Intervention Group A will be treated with SMT + Albumin + Midodrine (5mg thrice daily and will be increased every 3 days upto 15 mg thrice daily with target MAP (>75 mm and <90) and Group B with SMT + Albumin: 80grams/week for 2 weeks followed by 40gram/week + Placebo

Stopping ruleAdverse reaction to Albumin

* Cardiopulmonary compromise
* Allergic reaction

ELIGIBILITY:
Inclusion Criteria:

- Cirrhosis with refractory ascites

Exclusion Criteria:

- Recent Gastrointestinal bleeding within 7 days

* Systemic arterial hypertension (>160/90mmhg)
* Presence of hepatocellular carcinoma or portal vein thrombosis, Budd-chiari syndrome.
* Pregnancy
* No use of drugs affecting systemic hemodynamics 7 days prior to enrolment
* Patients with Cardiovascular disease (NYHA > II) or chronic obstructive pulmonary disease
* Refusal to participate
* Known or suspected hypersensitivity to albumin
* Prior TIPS
* Post liver or kidney transplantation
* Patients enrolled in other clinical trials
* Extrahepatic malignancy
* Patients on cardiac glycosides like digoxin, phenylephrine, ephedrine, thyroid hormones, ergot derivatives, salt retaining steroids like fludrocortisone, MAO inhibitors, alpha blockers metformin and ranitidine (known to have interactions with midodrine)
* Patients with intrinsic kidney disease, organ nephropathy and CKD stage 4 and
* MELD > 30 and extremely moribend patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-03-19 (Estimated); Study Completion 2022-03-19 (Estimated)

PRIMARY OUTCOMES:
Survival free of transplant and TIPS | 6 months

SECONDARY OUTCOMES:
Cumulative incidence of liver-related complications | 3 months
Cumulative incidence of liver-related complications | 6 months
Cumulative incidence of liver-related complications | 12 months
Survival free of liver transplant in both groups | 1 year
Survival free of TIPS in both groups | 1 year
Incidence of HRS-AKD, in both groups at 1 year | 1 year
Incidence of HRS-CKD in both groups at 1 year | 1 year
Incidence of HRS AKI in both groups at 1 year | 1 year
Cumulative frequency of large volume paracentesis | 3 months
Cumulative frequency of large volume paracentesis | 6 months
Cumulative frequency of large volume paracentesis | 12 months
Improvement in fraility | 3 months
  AS PER MAYO FRAITITY INDEX , FRAITILY IS CLASSIFIED AS PRE FRAIL, FRAIL AND ROBUST.
Improvement in fraility | 6 months
  AS PER MAYO FRAITITY INDEX , FRAITILY IS CLASSIFIED AS PRE FRAIL, FRAIL AND ROBUST.
Improvement in fraility | 12 months
  AS PER MAYO FRAITITY INDEX , FRAITILY IS CLASSIFIED AS PRE FRAIL, FRAIL AND ROBUST.
Survival free of TIPS | 6 months
Survival free of transplant at 6 months | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India